CLINICAL TRIAL: NCT06470022
Title: Randomized Comparison of Evolut FX Versus Sapien 3 Ultra Resilia. The Compare-TAVI 2 Trial
Brief Title: Comparison of Evolut FX Versus Sapien 3 Ultra Resilia.
Acronym: COMPARE-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Juhl Terkelsen (Other)
Collaborators: Department of Clinical Epidemiology, Aarhus University, DK-8200 Aarhus N, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Christian Juhl Terkelsen, Professor, MD, DmSc, PhD, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPARE-TAVI-2
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Randomized 1:1
Masking Description: The patient and operator cannot be blinded to allocated treatment. Most outcomes are registry based and randomization is not anticipated to impact outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Medtronic Evolut FX (Active Comparator): TAVI procedure performed with Medtronic Evolut FX
  Interventions: Device: Medtronic Evolut FX
- Edwards Sapien Ultra 3 Resilia (Active Comparator): TAVI procedure performed with Edwards Sapien Ultra 3 Resilia
  Interventions: Device: Edwards Sapien 3 Ultra Resilia

INTERVENTIONS:
Device: Medtronic Evolut FX — TAVI performed with Medtronic Evolut FX
  Arms: Medtronic Evolut FX
Device: Edwards Sapien 3 Ultra Resilia — TAVI performed with Edwards Sapien 3 Ultra Resilia
  Arms: Edwards Sapien Ultra 3 Resilia

SUMMARY:
To compare outcome in patients randomized to treatment with Evolut FX versus Sapien 3 Ultra Resilia.

DETAILED DESCRIPTION:
The purpose of the "Compare-TAVI" organization is to ensure a continuous comparison of the TAVI-valves implanted, and to monitor long-term valve performances.

Purpose of present study:

To compare outcome in patients randomized to treatment with Evolut FX versus Sapien 3 Ultra Resilia.

Hypotheses:

1. Evolut FX is non-inferior to Edwards Sapien 3 Resilia with regard to the combined endpoint (death, stroke, moderate/severe aortic regurgitation, moderate/severe valve deterioration) between the two valves being compared.
2. There is no difference between valves in secondary safety and efficacy endpoints (see below)
3. There is no difference in Aortic Regurgitation fraction (ARF) and Effective Orifice Area (EOA) measured by CMR (CMR-substudy, N=166)
4. There is no difference in EOA measured invasively during dobutamine stress (hemodynamic substudy, N=440).
5. There is no difference in occurrence of Hypoathenuated Leaflet Thickening (HALT) measured by CT (CT-substudy, N=778).

ELIGIBILITY:
Inclusion Criteria:

1. Patient more than 18 years of age.
2. Patient eligible for both Evolut FX and Edwards Sapien 3 Ultra Resilia according to a TAVI heart team conference.
3. The center experience for each of the valves considered should be more than 15 cases a year, and the treating physician should have implanted at least 15 of each valve used in the trial.
4. The center volume should be more than 75 cases a year.
5. The patient has given signed informed consent.
6. TAVI performed via the femoral artery.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1346 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality, stroke, moderate/major aortic regurgitation, moderate/severe THV deterioration | 1-year, 3-year, 5-year, 10-year
  The primary composite endpoint is at one-year, and a non-inferiority test is performed. See separate statistical analysis plan. Separate analyses of each component of the primary outcome will be presented, in accordance with the FDA guidelines and EMA guidelines, i.e. mortality, stroke, moderate/severe aortic regurgitation and moderate/severe THV deterioration to better understand their contribution to the primary endpoint. If non-inferiority is proven for the primary composite endpoint, a split alfa is used to test for superiority if possible (alfa=0.025) and to test secondary safety and efficacy endpoints (Total alfa=0.025 for these). The composite endpoint will be re-analyzed after 3-, 5- and 10-year as superiority analyses.

SECONDARY OUTCOMES:
TAVI-related complications | 7-days
  conversion to open surgery during implantation, unplanned use of cardiopulmonary support (CPS), coronary artery obstruction, ventricular septal perforation, mitral valve apparatus damage or dysfunction, cardiac tamponade / pericardial effusion resulting in pericardiocentesis, valve embolization, valve migration, need for TAVI-in-TAVI deployment, using VARC-3 criteria 10, or annulus rupture, aortic rupture/perforation, aortic dissection, or other shunts than VSD.
Proportion with successful implantation of the chosen valve. | 7-days
  This means no need for more than 1 TAVI valve, no change to another valve than planned during the procedure because it was impossible to implant the valve planned, and no conversion to surgery or procedure-related death.
SMART criteria for bioprosthetic valve dysfunction through 12 months | 1-year
  composed of the following components: (1) hemodynamic structural valve dysfunction, defined as aortic valve mean gradient ≥ 20 mmHg at any time up to the 12-month visit echo; (2) nonstructural valve dysfunction, defined as severe prosthesis-patient mismatch or ≥ moderate total aortic regurgitation at any time up to the 12-month visit echo; (3) clinical valve thrombosis; (4) endocarditis; or (5) aortic valve reintervention.
Pacemaker-implantation | 1-year
  New pace-maker implantation in pacemaker-naive patients.
Vascular and access-related complications (exploratory only) | 30-days
  Major vascular access site and access-related complications resulting in endovascular or open surgery using VARC-3 criteria
Bleeding and transfusion (exploratory only) | 30-days
  Major bleeding resulting in drop in hgb-level ≥1.86 mmol/l and/or erythrocyte transfusion ≥ 2 units, modified from BARC type 3-5 criteria
Endocarditis (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year
  According to VARC-3 criteria.
Reoperation (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year
  Transcatheter Aortic Valve Intervention, Surgical Aortic Valve Intervention or Balloon Angioplasty
Moderate/severe prosthesis-patient mismatch (exploratory only) | 30-day
  Effective Orifice Area (EOA)/body surface area ≤0.85 cm2/m2 if BMI<30 kg/cm2 or <=0.70 cm2/m2 if BMI>=30 kg/cm2., according to VARC-3 criteria.
Mean gradient (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year
  Aortic mean gradient, mmHg, as evaluated by Echocardiograpy Core-laboratory.
Pacemaker-implantation (exploratory only) | 30-day prior to TAVI, 30-day, 1-year, 3-year, 5-year, 10-year
  New pacemaker in pacemaker naive-patients.
Readmission for congestive heart failure (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year.
  Adjudicated. Only monitored until first confirmed case.
AMI (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year.
  Acute Myocardial Infarction. Adjudicated. Only monitored until first confirmed case.
Revascularization (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year.
  PCI (Percutaneous coronary intervention) CABG (Coronary Artery Bypass Grafting), not scheduled before TAVI
Atrial fibrillation (exploratory only) | 30-day, 1-year, 3-year, 5-year, 10-year.
  Newly diagnosed atrial fibrillation/flutter
Kidney injury (exploratory only) | 30-day
  Increase in renal creatinine level more than to ≥200% (AKIN stage 2-3, VARC-3 criteria) or resulting in dialysis (AKIN stage 4) according to VARC-3 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: christian J Terkelsen, Professor, Principal Investigator — Department of cardiology, Aarhus University Hospital, DK-8200 Aarhus N, Denmark
Locations (1):
- Department of cardiology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We are willing to collaborate in meta-analyses based on individual data where department of epidemiology, Aarhus University Hospital will be responsible for data-analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available now. Analytic will be made available when final statistical analyses performed.
Access Criteria: Contact primary investigator

DOCUMENTS (3):
  • Study Protocol (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/22/NCT06470022/Prot_004.pdf
  • Statistical Analysis Plan (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT06470022/SAP_005.pdf
  • Informed Consent Form (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT06470022/ICF_003.pdf